CLINICAL TRIAL: NCT01036646
Title: User Performance Evaluation of the INRatio® Prothrombin Time (PT) Monitoring System With a New INRatio Test Strip Designed for Low Sample Volume and Heparin Insensitivity
Acronym: ECLIPSE-02
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Other Study IDs: BSTE-0125
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Oral Anticoagulation
Keywords: Patients on stable OAT therapy for at least 3 months.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma specimens retained for reference method comparison.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BSTE-0125-Original Protocol
- BSTE-0125.a-Amended Protocol

SUMMARY:
This multi-center study is designed to evaluate the ability of intended lay users (patients on oral anticoagulation therapy, OAT, or their caregivers) to 1) operate the INRatio Prothrombin Time (PT) Monitoring System utilizing the INRatio test strip newly designed for low sample volume and heparin insensitivity, and 2) obtain accurate results for the quantitative determination of International Normalized Ratio (INR) when self-testing using fingerstick capillary blood. Patients will be trained by their healthcare provider using the instructions for use and product labeling provided. The accuracy of the patient INR results will be assessed by comparison to the INR results obtained by the site's trained healthcare professional using the same INRatio system (from a separate fingerstick collected from the same patient at the point-of-care), and with the INR results obtained on venous plasma obtained from the same patient and analyzed at a central laboratory with the Sysmex CA-560 System INR reference method.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older);
* Ability to read and speak English;
* Subjects on stable oral anticoagulation therapy with warfarin (at least 3 months);
* Target INR interval between 2.0 and 4.5
* Willing and able to provide written informed consent and comply with study procedures;

Exclusion Criteria:

* Hematocrit less than 25 or greater than 55%
* Lupus or antiphospholipid syndrome (APS)
* Already participated in this study
* A current INRatio PT Monitoring System User / Patient Self Tester

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from their primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Operate the INRatio Prothrombin Time (PT) Monitoring System utilizing the INRatio test strip newly designed for low sample volume and heparin insensitivity. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Loma Linda VA Hospital, Loma Linda, California
  - UC Davis Healthcare System, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - Fox Valley Cardiology, Aurora, Illinois